CLINICAL TRIAL: NCT04943055
Title: Multi-center Clinical Study of Low Temperature Plasma Ablation Combined With Lacrimal Duct Catheterization in the Treatment of Lacrimal Duct Obstructive Diseases
Brief Title: Low Temperature Plasma Ablation Combined Lacrimal Duct Catheterization in the Treatment of Lacrimal Duct Obstructive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-151
Record Dates: First submitted 2021-06-10; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Lacrimal Duct Obstruction
Keywords: Lacrimal Duct Obstruction; Low temperature plasma ablation
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low temperature plasma ablation with lacrimal duct catheterization (Experimental): The experimental group received low temperature plasma lacrimal duct obstruction ablation combined with lacrimal duct catheterization
  Interventions: Procedure: Low temperature plasma lacrimal duct obstruction ablation combined with lacrimal duct catheterization
- YAG lacrimal duct laser combined with lacrimal duct catheter (Placebo Comparator): Control group received YAG lacrimal duct laser combined with lacrimal duct catheterization
  Interventions: Procedure: YAG lacrimal duct laser combined with lacrimal duct catheter

INTERVENTIONS:
Procedure: Low temperature plasma lacrimal duct obstruction ablation combined with lacrimal duct catheterization — The operation used a tear point dilator to expand the patient's upper and lower tear points, YAG laser/low-temperature plasma knife was used to clear the obstructed site of the patient, and normal saline was used to rinse to ensure the patency of the lacrimal passage. The silicone lacrimal duct drainage tube was selected to put the lacrimal duct drainage tube in the upper and lower lacrimal dots of the patient, and the metal probe was removed after using a crochet, and the drainage tube was moderately pulled upward from the center of the upper and lower lacrimal dots to facilitate the smooth passage of the drainage tube through the whole lacrimal duct and achieve the purpose of dredging the blocked site again. Adjust the length of the drainage tube in the nasal vestibule and leave it in the nasal cavity.
  Arms: Low temperature plasma ablation with lacrimal duct catheterization
Procedure: YAG lacrimal duct laser combined with lacrimal duct catheter — The operation used a tear point dilator to expand the patient's upper and lower tear points, YAG laser/low-temperature plasma knife was used to clear the obstructed site of the patient, and normal saline was used to rinse to ensure the patency of the lacrimal passage. The silicone lacrimal duct drainage tube was selected to put the lacrimal duct drainage tube in the upper and lower lacrimal dots of the patient, and the metal probe was removed after using a crochet, and the drainage tube was moderately pulled upward from the center of the upper and lower lacrimal dots to facilitate the smooth passage of the drainage tube through the whole lacrimal duct and achieve the purpose of dredging the blocked site again. Adjust the length of the drainage tube in the nasal vestibule and leave it in the nasal cavity.
  Arms: YAG lacrimal duct laser combined with lacrimal duct catheter

SUMMARY:
To compare the clinical effects of low temperature plasma ablation combined with lacrimal duct catheterization and YAG lacrimal duct laser combined with lacrimal duct catheterization in the treatment of lacrimal duct obstruction

DETAILED DESCRIPTION:
Low-temperature plasma technology has developed rapidly in recent decades and is now widely used in ophthalmology, otolaryngology, orthopedics, urology and other fields .The low-temperature plasma surgery system relies on a 100kHz radio frequency electric field to excite normal saline (0.9% NaCl) to generate plasma energy, and relies on a 50-100 μm plasma layer generated at the front of the plasma knife to perform precise cutting, ablation and hemostaxy. But the application of this technique in the field of lacrimal duct still needs the accumulation of clinical experience.This study was aimed to compare the clinical effects of low temperature plasma ablation combined with lacrimal duct catheterization and YAG lacrimal duct laser combined with lacrimal duct catheterization in the treatment of lacrimal duct obstruction

ELIGIBILITY:
Inclusion Criteria:

* ① sign the informed consent for this study Voluntarily

  * ≥18 years old and < 70 years old (3) Single lacrimal tract obstruction was included in the study

    * no purulent secretion of lacrimal passage

Exclusion Criteria:

* Patients who meet any of the following criteria will not be eligible for inclusion in this study:

  * Have a history of lacrimal duct surgery, including lacrimal duct catheterization, laser lacrimal duct plasty, etc

    * Have a history of allergy to hormones and antibiotics

      * congenital lacrimal duct malformation

        * nasal trauma and deformation ⑤ Patients with severe abnormal liver and kidney function and cardiovascular and cerebrovascular diseases In addition to lacrimal duct obstruction, there are other ophthalmic diseases ⑦ Exclude diabetes

          * Exclusion of pregnancy, lactation women ⑨ Not willing to participate in research

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2023-07-07 (Estimated); Study Completion 2023-08-07 (Estimated)

PRIMARY OUTCOMES:
Change between 1 week, 1, 2, 3 months and 6 months postoperatively of degree of watering | Postoperatively 1 week, 1, 2, 3 months, 6 months
  The degree of watering was evaluated and classified according to the following clinical symptoms: 1 = no epiphora, 2 = minimal epiphora outdoors but only with wind or cold, 3 = troublesome epiphora outdoors but not indoors, 4 = epiphora indoors and outdoors

SECONDARY OUTCOMES:
Change between 1 week, 1, 2, 3 months and 6 months postoperatively of intraoperative complications | Postoperatively 1 week, 1, 2, 3 months, 6 months
  The complications of laser or plasma treatment involve abnormal tear secretion, acute and chronic purulent dacryocystitis, sepsis, false passage formation, epistaxis, and subcutaneous emphysema
Change between 1 week, 1, 2, 3 months and 6 months postoperatively of pain score | Postoperatively 1 week, 1, 2, 3 months, 6 months
  The VAS pain grade was recorded on a 0-10 scale, with 0 being no pain and 10 being the most intense pain

CONTACTS AND LOCATIONS:
Overall Officials: lin lin, Study Chair — Second Affiliated Hospital of Zhejiang University Hospital
Locations (1):
- Second Affiliated Hospital of Zhejiang University Hospital, Hangzhou, China